CLINICAL TRIAL: NCT03147976
Title: A Phase 2 Study of AMG 337 in Subjects With Advanced or Metastatic Solid Tumors That Overexpress Mesenchymal Epithelial Transition (MET) or Harbor MET Exon 14 Skipping (METex14del) Mutations
Brief Title: QUILT-3.036: AMG 337 in Subjects With Advanced or Metastatic Solid Tumors
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Enrollment not initiated
Sponsor: NantPharma, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QUILT-3.036
Record Dates: First submitted 2017-05-08; First posted 2017-05-10 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2018-08

CONDITIONS: Solid Tumor
MeSH Terms: interventions — AMG 337

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AMG 337 (Experimental): AMG 337 in subjects with advanced or metastatic solid tumors that overexpress MET or harbor METex14del mutations
  Interventions: Drug: AMG 337

INTERVENTIONS:
Drug: AMG 337 — 6-{(1R)-1-[8-fluoro-6-(1-methyl-1H-pyrazol-4- yl)[1,2,4]triazolo[4,3-a]pyridin-3-yl]ethyl}-3-(2- methoxyethoxy)-1,6-naphthyridin-5(6H)-one•hydrate (1:1)

SUMMARY:
This is a phase 2 study of AMG 337 in subjects with advanced or metastatic solid tumors that overexpress MET or harbor METex14del mutations resulting in MET exon 14 skipping.

DETAILED DESCRIPTION:
This is a phase 2, two-cohort, single-arm open-label study that will assess the efficacy of AMG 337 based on ORR in subjects with advanced or metastatic solid tumors that overexpress MET or harbor METex14del mutations resulting in MET exon 14 skipping. MET overexpression will be determined by quantitative proteomics with mass spectrometry. METex14del mutations resulting in MET exon 14 skipping will be determined by DNA sequencing and confirmed with RNA sequencing. Subjects will be enrolled as follows:

* Cohort 1: Subjects with advanced or metastatic solid tumors that overexpress MET
* Cohort 2: Subjects with advanced or metastatic solid tumors that harbor METex14del mutations Simon's two-stage optimal design will be utilized separately for each cohort to assess the primary efficacy endpoint ORR. The null hypothesis of Simon's two-stage design states that the ORR will be ≤ 10% (poor response) and will be tested against a one-sided alternative.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and provide a signed informed consent that fulfills the relevant Institutional Review Board (IRB) or Independent Ethics Committee (IEC) guidelines.
2. Able to attend required study visits and return for adequate follow-up, as required by this protocol.
3. Able to self-administer AMG 337 as a whole capsule by mouth every day.
4. Age ≥ 16 years old.
5. Histologically confirmed, unresectable locally advanced or metastatic solid tumor that overexpresses tumor MET (determined by quantitative proteomics with mass spectrometry [cohort 1]) or harbor METex14del mutations resulting in MET exon 14 skipping (as determined by DNA sequencing and confirmed with RNA sequencing [cohort 2]).
6. Have measurable disease evaluable in accordance with RECIST Version 1.1.
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
8. Must have a recent formalin-fixed paraffin-embedded (FFPE) tumor biopsy specimen that was obtained following the conclusion of the most recent anticancer treatment. If a historic specimen is not available, the subject must be willing to undergo a biopsy during the screening period, if considered safe by the Investigator. If safety concerns preclude collection of a biopsy during the screening period, a tumor biopsy specimen collected prior to the conclusion of the most recent anticancer treatment may be used.
9. Must be willing to undergo a biopsy during the treatment period, if considered safe by the investigator.
10. Ability to attend required study visits and return for adequate follow-up, as required by this protocol.
11. Hematologic function, as follows:

    1. Absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L.
    2. Platelet count ≥ 50 × 10^9/L.
    3. Hemoglobin > 8 g/dL.
    4. Prothrombin time (PT) or partial thromboplastin time (PTT) < 1.5 × upper limit of normal (ULN), except for subjects on anticoagulation therapy for venous thromboembolism.
12. Renal function, as follows:

    a. Calculated creatinine clearance > 30 mL/min.
13. Hepatic function, as follows:

    1. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2.5 × ULN and total bilirubin < 1.5 × ULN.
    2. Alkaline phosphatase (ALP) < 2 × ULN (≤ 5 × ULN if bone or liver metastases are present).
14. Agreement to practice effective contraception (both male and female subjects, if the risk of conception exists).

Exclusion Criteria:

1. Assessed by the investigator to be unable or unwilling to comply with the requirements of the protocol.
2. Inability to attend required study visits and return for adequate follow-up, as required for this protocol.
3. Known hypersensitivity to any component of the study medication(s).
4. Women who are nursing, pregnant, or planning to become pregnant during the duration of the study.
5. Current diagnosis of sporadic or hereditary renal cell carcinoma.
6. Current diagnosis or history of a second neoplasm, except the following:

   a. Adequately treated non-melanoma skin cancer, curatively treated in situ disease, or other solid tumors curatively treated with no evidence of disease for ≥ 2 years.
7. Subjects with tumors with ALK-positive rearrangement who received prior treatment with crizotinib.
8. History of bleeding diathesis.
9. Uncontrolled hypertension (systolic > 160 mmHg and/or diastolic > 100 mmHg) or clinically significant cardiovascular disease, cerebrovascular accident/stroke, or myocardial infarction within 6 months before study day 1; unstable angina; congestive heart failure of New York Heart Association grade 2 or higher; or serious cardiac arrhythmia requiring medication.
10. Baseline ECG Fridericia's formula (QTcF) > 470 ms.
11. Active infection requiring IV antibiotics within 2 weeks before study day 1.
12. Significant gastrointestinal disorder (eg, Crohn's disease, ulcerative colitis, extensive gastrointestinal resection) that in the opinion of the investigator may influence drug absorption.
13. Positive result of screening test for human immunodeficiency virus (HIV).
14. Evidence of acute hepatitis B and C. Subjects with chronic hepatitis B or C are eligible if their condition is stable and, in the opinion of the investigator, would not pose a risk to subject safety.
15. Toxicities from prior anti-tumor therapy not resolved to CTCAE Version 4.03 grade 0 or 1.

    a. Grade 2 toxicities from prior antitumor therapy that are considered irreversible (defined as having been present or stable for > 4 weeks), such as stable grade 2 peripheral neuropathy or ifosfamide-related proteinuria, may be allowed if they are not otherwise described in the exclusion criteria.
16. Participation in this study or in an investigational study and/or procedure with any molecularly targeted agents reported to inhibit MET within 14 days before study day 1.
17. Antitumor therapy, including chemotherapy, antibody therapy, retinoid therapy, or other investigational therapy, within 14 days before study day 1.
18. Therapeutic or palliative radiation therapy within 14 days before study day 1.
19. Major surgery within 28 days before study day 1.
20. Any comorbidity that in the opinion of the investigator may increase the risk of toxicity.
21. Concurrent or prior use of a strong CYP3A4 inhibitor within 14 days before study day 1, including the following: ketoconazole, itraconazole, clarithromycin, indinavir, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, and voriconazole.
22. Concurrent or prior ingestion of grapefruit, grapefruit products, or other foods known to inhibit CYP3A4 within 7 days before study day 1.
23. Concurrent or prior use of strong CYP3A4 inducers within 28 days before study day 1, including the following: phenytoin, carbamazepine, rifampin, rifabutin, rifapentin, phenobarbital, and the herbal supplement St. John's Wort.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2019-08-23 (Actual); Study Completion 2019-08-23 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 1 year
  Confirmed ORR (confirmed complete response (CR) or partial response (PR)) will be evaluated in accordance with RECIST Version 1.1.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (Safety And Tolerability) | 1 year
  To evaluate the safety of AMG 337 based on grade 3 or 4 non-hematologic toxicity
Progression-free Survival (PFS) | 1 year
  To determine PFS, evaluated in accordance with RECIST Version 1.1.
Overall Survival (OS) | 1 year
  To determine OS, defined as the time from the date of the first administration of therapy to the date of death.
Duration of Response (DOR) | 1 year
  To determine the duration of response, measured by RECIST Version 1.1.
Disease Control Rate (DCR) | 4 months
  To determine disease control rate (confirmed CR, PR, or stable disease [SD]) lasting for at least 4 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Chan Soon-Shiong Institute for Medicine, El Segundo, California, United States

IPD SHARING:
Plan to Share IPD: No